CLINICAL TRIAL: NCT06589219
Title: A Phase 1/1B Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Nebulized CMR316 in Healthy Volunteers and Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Study to Assess CMR316 in Healthy Volunteers and Patients With Idiopathic Pulmonary Fibrosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Calibr, a division of Scripps Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBR-CMR316-3001
Record Dates: First submitted 2024-08-19; First posted 2024-09-19 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Fibroses, Idiopathic
Keywords: Pulmonary; IPF; Inhaled therapy
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: Part 1 Cohorts 1-4: double-blind, assess single ascending doses (SAD) of nebulized CMR316. Cohort 5: open label, single dose (at a dose previously determined to be safe) & incl. lung sample collection via bronchoscopy for PK & PD.
  Part 2: double blind, assess multiple ascending dose (MAD) cohorts of CMR316 administered once weekly for 4 weeks. If further PK/PD data from lung samples is required to determine appropriate RP2D then a sub-group of open-label participants who will undergo bronchoscopies may be enrolled to any or all MAD cohorts.
  Parts 1 &2 are not required to be conducted entirely sequentially if justified by PK & safety obtained. The first MAD cohort will not start until data are available from SAD Cohort 3 & dosing for each MAD cohort will not exceed a dose level previously deemed safe in a SAD cohort. Part 3: IPF patients, will not start until data are available and reviewed from Parts 1 & 2 and will not exceed a dose level previously deemed safe in a SAD/MAD cohort.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The majority of this study will be conducted double-blind; treatment assignment will not be known to the subjects, the Sponsor (with exception of an unblinded bioanalytical specialist who will review PK and PD and blind data for presentation to blinded team) and staff involved in the clinical evaluation of the subjects and the analysis of data. The randomization schedule and disclosure envelopes will be generated by an unblinded statistical team. The unblinded statistical team will not be involved in decisions relating to populations for analysis prior to unblinding. Prior to database lock and unblinding, all original randomization materials will be held by the unblinded statistical team. There may be instances where interim data has the potential to reveal treatment. In these cases, every effort will be made by the unblinded bioanalytical specialist to maintain blinding by appropriate presentation of data to the study team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part 1 SAD CMR316 (Active Comparator): Single ascending dose, nebulized administration of CMR316
  Interventions: Drug: CMR316
- Part 1 SAD Placebo (Placebo Comparator): Single ascending dose, nebulized administration of matching placebo
  Interventions: Drug: Placebo
- Part 2 MAD CMR316 (Active Comparator): Multiple ascending dose, nebulized administration of CMR316 once weekly for 4 weeks
  Interventions: Drug: CMR316
- Part 2 MAD Placebo (Placebo Comparator): Multiple ascending dose, nebulized administration of matching placebo once weekly for 4 weeks
  Interventions: Drug: Placebo
- Part 3 IPF Patients (Experimental): Open-label, nebulized administration of CMR316 once weekly for 4 weeks for patients with IPF
  Interventions: Drug: CMR316

INTERVENTIONS:
Drug: CMR316 — CMR316 administered via nebulization at single or multiple dose(s) assigned by cohort
  Arms: Part 1 SAD CMR316; Part 2 MAD CMR316; Part 3 IPF Patients
Drug: Placebo — Placebo administered via nebulization at single or multiple dose(s) to match CMR316 administration
  Arms: Part 1 SAD Placebo; Part 2 MAD Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics single and multiple inhaled doses of CMR316 in healthy volunteers and patients with Idiopathic Pulmonary Fibrosis (IPF).

DETAILED DESCRIPTION:
This is a 3-part, single-center study; Part 1 will evaluate single ascending doses (SAD) and Part 2 will evaluate multiple ascending doses (MAD; once weekly dosing for 4 weeks) of nebulized CMR316 or placebo in healthy male and female subjects. Part 3 will assess multiple doses (once weekly dosing for 4 weeks) of nebulized CMR316 (open-label) in subjects with IPF.

ELIGIBILITY:
Inclusion Criteria: Part 1 & 2

* Healthy men or non-pregnant, non-lactating healthy women of non-childbearing potential, 18-60 years of age.
* Must agree to use a highly effective method of contraception.
* Body Mass Index (BMI) 18-33 kg/m2 as measured at screening.
* Weight ≤100 kg at screening.
* Normal lung function, defined as: FVC and FEV1 > 80% predicted (based on age, height, race, sex, SaO2 > 95% on room air.
* Heart rate between 50 and 90 beats per minute (BPM).
* Good state of health (mentally and physically) as indicated by a comprehensive clinical assessment (detailed medical history and a complete physical examination) and screening safety procedures.

Inclusion Criteria: Part 3

* Diagnosis of IPF by American Thoracic Society/ERS (European Respiratory Society)/JRS (Japanese Respiratory Society)/ALAT (Latin America Thoracic Society) 2011 criteria within five years prior to consent.
* Men or non-pregnant, non-lactating women of non-childbearing potential.
* Age ≥ 40 years.
* Mild to moderate IPF as defined by predicted FVC ≥ 55% of normal and predicted DLCO > 40% of normal at Screening.
* Subjects receiving oral pirfenidone or nintedanib for treatment of IPF may participate if they have been on treatment with a stable, well-tolerated dose (as determined by the investigator), for at least 8 weeks prior to consent with no changes to therapy dose and schedule anticipated during the course of study participation.
* Must be able to understand a written informed consent, which must be obtained prior to any study procedures.
* Must be willing and able to comply with all study requirements

Exclusion Criteria: Part 1 & 2

* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients.
* Presence or history of clinically significant hypersensitivity (e.g., anaphylaxis, angioedema, Stevens-Johnson syndrome) or allergy as judged by the investigator. Subjects with a history of seasonal rhinitis (hay fever) or childhood asthma may participate if these conditions are not active or expected to be active during the subject's participation.
* History of clinically significant cardiovascular, skin, renal, hepatic, respiratory or gastrointestinal disease (except cholecystectomy), neurological or psychiatric disorder, illness/infection/hospitalization, or surgical procedure within 30 days prior to first dose of study drug. Subjects with a history of pancreatitis, heart failure, acute renal failure, bullous pemphigoid, or severe and disabling arthritis, conditions associated with postmarketing safety reports of oral gliptins, are excluded.
* Have poor venous access that limits phlebotomy.
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and bilirubin above upper limit of normal (elevated bilirubin in subject's with Gilbert Syndrome is allowed) or other clinically significant abnormal clinical chemistry, hematology, or urinalysis as judged by the investigator.
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), or human immunodeficiency virus (HIV) antibody results.
* Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance (CLcr) of <90 mL/min using the 2021 Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation (Appendix 1: CKD-EPI Equation).
* Subjects with a corrected QT interval by Fredericia (QTcF) of >450 msec at screening or first admission.
* Positive highly sensitive serum pregnancy test at screening or highly sensitive urine pregnancy test at first admission. Those who are pregnant or lactating will be excluded.
* Subjects who have received any investigational medicinal product (IMP) in a clinical research study within 5 half-lives or within 30 days prior to first dose (whichever is longer).
* Subjects who have previously been administered IMP in this study. Subjects who have taken part in Part 1 are not permitted to take part in Part 2.
* Subjects who have taken, any over-the-counter drug or herbal remedies in the 15 days prior to first IMP administration. Subjects taking prescribed medication in the 90 days prior to first IMP administration. Subjects taking up to 4 g per day of acetaminophen may participate if discontinued at least 15 days prior to first IMP administration. Subjects taking DPP4 inhibitors are prohibited. Subjects taking strong CYP3A inhibitors are prohibited.
* History of any substance use disorder or alcohol use disorder in the past 2 years, as based on the diagnostic criteria in the Diagnostic and Statistical Manual Fifth Edition (DSM-5).
* Regular alcohol consumption in men >21 units per week and women >14 units per week (1 unit = 12 oz 1 bottle/can of beer, 1 oz 40% spirit, or 5 oz glass of wine).
* A confirmed positive alcohol breath test at screening or first admission.
* Current smokers and those who have a smoking history of ≥ 10 pack-years. A confirmed positive urine cotinine test at screening or first admission.
* Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months.
* Positive test result for common drugs of abuse on screening and first admission.
* Men with pregnant or lactating partners.
* Donation of a unit of blood (about 500 mL) within 2 months or donation of plasma within 7 days prior to first dose of study medication.
* Subjects who are, or are immediate family members of, a study site or Sponsor employee.
* Active respiratory infection requiring treatment with antibiotics within 4 weeks prior to signing of ICF.
* Lack of suitability for participation in the trial, for any reason, as judged by the Investigator.

Exclusion Criteria: Part 3

* Clinically significant deterioration between screening and Day 1.
* Use of any investigational drugs within 30 days or 5 half-lives prior to consent, whichever is longer.
* Serious adverse reaction or serious hypersensitivity to any DPP4 inhibitor (e.g., saxagliptin, sitagliptin) or the formulation excipients.
* Use of supplemental oxygen for resting hypoxemia.
* Evidence of significant renal impairment at screening, defined in this protocol as an estimated creatinine clearance (CLcr) of <50 mL/min using the CKD-EPI equation. Patients with renal insufficiency Clcr ≥ 50 mL/min with stable renal function (per clinical discretion, recommend based on average documented clinical chemistry values for at least 6 months) may participate.
* History of clinically significant and uncontrolled medical illness or clinically significant abnormal clinical chemistry, hematology, or urinalysis that represents a meaningful risk to the subject during this trial, as judged by the Investigator (e.g., heart failure).
* Subjects with a corrected QT interval by Fredericia (QTcF) of >450 msec at screening.
* Life expectancy < one year.
* Subject listed for lung transplant.
* Hospitalization or serious illness (as determined by the investigator) within the 3 months prior to consent.
* Alternative diagnoses that could lead to pulmonary fibrosis such as exposure to drugs, radiation, asbestos.
* Connective tissue disease that can lead to pulmonary fibrosis such as scleroderma or rheumatoid arthritis.
* Presence of clinically active, medically diagnosed asthma, chronic obstructive pulmonary disease, or active infection.
* Lack of suitability for participation in the trial, for any reason, as judged by the Investigator.
* History of severe hepatic impairment or AST or ALT greater than 3 times the upper limit of normal at screening.
* The use of required concomitant medications that represents a significant risk to produce an adverse drug interaction with CMR316, assessed by the investigator (in consultation with sponsor and sponsor's medical monitor). Specifically, subjects with Type 1 and Type 2 diabetes are excluded.
* Smoking within a year prior to consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | Part 1: Day 1 through Day 5; Part 2: Day 1 through Day 26; Part 3: Day 1 through Day 26
  Adverse events will be analyzed for severity and potential relationship to CMR316 to determine safety and tolerability of CMR316
Number of participants with clinically significant abnormal physical exam and vital signs | Part 1: Day 1 through Day 5; Part 2: Day 1 through Day 26; Part 3: Day 1 through Day 26
  Vital signs will include evaluation of systolic and/or diastolic blood pressure (mmHg), heart rate (beats/min), temperature (Celsius), and respiratory rate (breaths/minute).
Number of patients with reduced pulmonary function | Part 1: Day 1 through Day 5; Part 2: Day 1 through Day 26; Part 3: Day 1 through Day 26
  Pulse oximeter will analyze oxygen saturation, spirometry will include evaluation of FEV1, FVC, and FEV1/FVC, and DLCO
Number of participants with abnormal electrocardiogram readings | Part 1: Day 1 through Day 5; Part 2: Day 1 through Day 26; Part 3: Day 1 through Day 26
  Electrocardiogram will include an evaluation of QTcF interval, ventricular rate, PR interval, QRS duration and QRS axis
Number of participants with clinically significant abnormal laboratory test results | Part 1: Day 1 through Day 5; Part 2: Day 1 through Day 26; Part 3: Day 1 through Day 26
  Results outside of laboratory defined normal ranges will be analyzed for clinical significance and used to determine safety and tolerability of CMR316

SECONDARY OUTCOMES:
Assess pharmacokinetics, AUC, as available | Part 1: Day 1 through Day 15; Part 2: Day 1 through Day 36; Part 3: Day 1 through Day 36
  Area under the concentration-time curve (AUC) from time of administration
Assess pharmacokinetics, Cmax, as available | Part 1: Day 1 through Day 15; Part 2: Day 1 through Day 36; Part 3: Day 1 through Day 36
  Maximum drug concentration observed
Assess pharmacodynamics, characterize enzymatic activity | Part 1: Day 1 though Day 8; Part 2: Day 1 through Day 29; Part 3: Day 1 through Day 29
  Change from pre-dose baseline and % inhibition in enzymatic activity

CONTACTS AND LOCATIONS:
Overall Officials: Chan Beals, MD, PhD, Principal Investigator — Calibr-Skaggs Institute for Innovative Medicines
Locations (1):
- Fraunhofer Institute for Toxicology and Experimental Medicine ITEM, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No